CLINICAL TRIAL: NCT03439462
Title: A Phase 1/2 Multi-center Investigation of ABI-009 (Nab-rapamycin) in Combination With FOLFOX and Bevacizumab as First-line Therapy in Patients With Advanced or Metastatic Colorectal Cancer
Brief Title: Nab-Sirolimus in Combination With FOLFOX & BEV as 1st Line Therapy in Patients With Advanced or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aadi Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COLO-007
Record Dates: First submitted 2018-02-08; First posted 2018-02-20 (Actual); Results first posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- nab-sirolimus (also known as ABI-009, nab-rapamycin, albumin-bound rapamycin) (Experimental): Single arm, open-label, multi-institutional study to identify the RP2D and determine the efficacy and safety profile of nab-sirolimus administered as first-line therapy in combination with mFOLFOX6 and bevacizumab in patients with metastatic CRC.
  Interventions: Drug: nab-sirolimus

INTERVENTIONS:
Drug: nab-sirolimus — nab-sirolimus combined with mFOLFOX6 + bevacizumab
  Other Names: bevacizumab; mFOLFOX6

SUMMARY:
A phase 1/2 multi-center investigation of nab-sirolimus (also known as ABI-009, nab-rapamycin) in combination with mFOLFOX6 and Bevacizumab as first-line therapy in patients with metastatic colorectal cancer

DETAILED DESCRIPTION:
This study is a prospective phase 1/2, single arm, open-label, multi-institutional study to identify the RP2D and determine the efficacy and safety profile of nab-sirolimus administered as first-line therapy in combination with mFOLFOX6 and bevacizumab in patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed advanced or metastatic colorectal cancers for whom chemotherapy is indicated.
2. Patients must not have had prior chemotherapy for advanced or metastatic disease. Patients could have received adjuvant chemotherapy or adjuvant chemo-radiotherapy.
3. Patients must have at least 1 measurable site of disease according to RECIST v1.1 that has not been previously irradiated. If the patient has had previous radiation to the marker lesion(s), there must be radiological evidence of progression since the radiation.
4. Eligible patients, 18 years or older, with Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
5. Patients must not have been previously treated with an mTOR inhibitor.
6. Adequate liver function:

   1. Total bilirubin ≤1.5 x upper limit of normal (ULN) mg/dL
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x ULN (<5 x ULN if the patient has liver metastases).
7. Adequate renal function:

   a. Serum creatinine ≤2 x ULN or creatinine clearance >50 cc/hr (Cockroft-Gault).
8. Adequate biological parameters:

   1. Absolute neutrophil count (ANC) ≥1.5 × 109/L
   2. Platelet count ≥100,000/mm3 (100 × 109/L)
   3. Hemoglobin ≥9 g/dL.
9. Fasting serum triglyceride ≤300 mg/dL; fasting serum cholesterol ≤350 mg/dL.
10. INR and PTT <1.5 x ULN (anticoagulation is allowed if target INR <1.5 on a stable dose of warfarin or on a stable dose of LMW heparin for >2 weeks at time of enrollment).
11. Minimum of 4 weeks since any major surgery, completion of radiation, or completion of all prior systemic anticancer therapy, and ≥6 months since adjuvant FOLFOX therapy (adequately recovered from the acute toxicities of any prior therapy, including neuropathy should be grade ≤1).
12. Male or non-pregnant and non-breast feeding female:

    * Females of child-bearing potential must agree to use effective contraception without interruption from 28 days prior to starting IP throughout 3 months after last dose of IP and have a negative serum pregnancy test (β -hCG) result at screening and agree to ongoing pregnancy testing during the course of the study, and after the end of study treatment. A second form of birth control is required even if she has had a tubal ligation.
    * Male patients must practice abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study and throughout 3 months after last dose of IP. A second form of birth control is required even if he has undergone a successful vasectomy.
13. Life expectancy of >3 months, as determined by the investigator.
14. Ability to understand and sign informed consent.
15. Willingness and ability to comply with scheduled visits, laboratory tests, and other study procedures.

Exclusion Criteria:

1. History of severe and uncontrolled allergic reactions to bevacizumab
2. Prior treatment with FOLFOX or bevacizumab within the preceding 4 weeks
3. Patients currently receiving or have received anticancer therapies within 4 weeks of the start of study treatment (including chemotherapy, radiation therapy, antibody based therapy, etc.)
4. Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study
5. Chronic treatment with systemic steroids or another immunosuppressive agent; topical or inhaled corticosteroids are allowed
6. Recent infection requiring systemic anti-infective treatment that was completed ≤14 days prior to enrollment (with the exception of uncomplicated urinary tract infection or upper respiratory tract infection).
7. Patients who have any severe and/or uncontrolled medical or psychiatric conditions or other conditions that could affect their participation including:

   1. Known active uncontrolled or symptomatic central nervous system (CNS) metastases. A patient with controlled and asymptomatic CNS metastases may participate in this study. As such, the patient must have completed any prior treatment for CNS metastases ≥28 days (including radiotherapy and/or surgery) prior to start of treatment in this study and should not be receiving chronic corticosteroid therapy for the CNS metastases.
   2. Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6 months prior to first study treatment, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
   3. Pre-existing severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or O2 saturation that is 88% or less at rest on room air (Note: spirometry and PFTs not required to be performed unless clinically indicated).
   4. Uncontrolled diabetes as defined by fasting serum glucose >1.5x ULN or by HbA1c >8% despite adequate therapy.
   5. Any active (acute or chronic) or uncontrolled infection/ disorders.
   6. Nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy. Note, controlled non-melanoma skin cancers, carcinoma in situ of the cervix, resected incidental prostate cancer, or other adequately treated carcinoma-in-situ may be eligible, after documented discussion with the sponsor / medical monitor.
   7. Known liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C).
8. Patients with history of interstitial lung disease and/or pneumonitis, or pulmonary hypertension.
9. A known history of HIV seropositivity.
10. Active Hepatitis B or Hepatitis C. Note: A detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients. HBV DNA and HCV RNA PCR testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection.
11. Patients with an active bleeding diathesis or on oral anti-vitamin K medication (except low dose Coumadin).
12. Use of strong inhibitors and inducers of CYP3A4 within the 14 days prior to receiving the first dose of ABI-009. Additionally, use of any known CYP3A4 substrates with narrow therapeutic window (such as fentanyl, alfentanil, astemizole, cisapride, dihydroergotamine, pimozide, quinidine, terfanide) within the 14 days prior to receiving the first dose of ABI-009.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Atlantic Health System/Morristown Medical Center, Morristown, New Jersey
  - Baylor Scott and White University Medical Center, Dallas, Texas
  - Seattle Cancer Care Alliance/University of Washington Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Cohort 1: Nab-Sirolimus 30 mg/m2 qw3/4: Dose / Schedule Cohort 1:
  nab-Sirolimus: 30 mg/m2 weekly on Days 1, 8, and 15 (28-day cycle) by IV
  Modified FOLFOX6 regimen: oxaliplatin 85 mg/m2 IV with LV 400 mg/m2 IV plus FU 400 mg/m2 IV bolus and 2,400 mg/m2 continuous infusion over 46 hours every 2 weeks
  Bevacizumab: 5 mg/kg IV every 2 weeks
- Cohort 2: Nab-Sirolimus 20 mg/m2 qw3/4: Dose / Schedule Cohort 2:
  nab-Sirolimus: 20 mg/m2 weekly on Days 1, 8, and 15 (28-day cycle) by IV
  Modified FOLFOX6 regimen: oxaliplatin 85 mg/m2 IV with LV 400 mg/m2 IV over 2 hours plus FU 400 mg/m2 IV bolus and 2,400 mg/m2 continuous infusion over 46 hours every 2 weeks
  Bevacizumab: 5 mg/kg IV every 2 weeks
- Cohort 3: Nab-Sirolimus 20 mg/m2 qw2/4: Dose / Schedule Cohort 3 (Recommended Phase 2 Dose, RP2D):
  nab-Sirolimus: 20 mg/m2 every 2 weeks (28-day cycle) by IV
  Modified FOLFOX6 regimen: oxaliplatin 85 mg/m2 IV with LV 400 mg/m2 IV over 2 hours plus FU 400 mg/m2 IV bolus and 2,400 mg/m2 continuous infusion over 46 hours every 2 weeks
  Bevacizumab: 5 mg/kg IV every 2 weeks
Period: Overall Study
Arm/Group | Dose Cohort 1: Nab-Sirolimus 30 mg/m2 qw3/4 | Cohort 2: Nab-Sirolimus 20 mg/m2 qw3/4 | Cohort 3: Nab-Sirolimus 20 mg/m2 qw2/4
Started | 6 | 10 | 44
Completed | 6 | 10 | 44
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set includes all treated patients
Groups:
- Cohort 1: Nab-Sirolimus 30 mg/m2 qw3/4: Dose /Schedule Cohort 1:
  nab-Sirolimus: 30 mg/m2 weekly on Days 1, 8, and 15 (28-day cycle) by IV
  Modified FOLFOX6 regimen: oxaliplatin 85 mg/m2 IV with LV 400 mg/m2 IV over 2 hours plus FU 400 mg/m2 IV bolus and 2,400 mg/m2 continuous infusion over 46 hours every 2 weeks
  Bevacizumab: 5 mg/kg IV every 2 weeks
- Cohort 1: Nab-Sirolimus 20 mg/m2 qw3/4: Dose /Schedule Cohort 2:
  nab-Sirolimus: 20 mg/m2 weekly on Days 1, 8, and 15 (28-day cycle) by IV
  Modified FOLFOX6 regimen: oxaliplatin 85 mg/m2 IV with LV 400 mg/m2 IV over 2 hours plus FU 400 mg/m2 IV bolus and 2,400 mg/m2 continuous infusion over 46 hours every 2 weeks.
  Bevacizumab: 5 mg/kg IV every 2 weeks
- Cohort 2: Nab-Sirolimus 20 mg/m2 qw2/4: Dose /Schedule Cohort 3: (Recommended Phase 2 Dose, RP2D):
  nab-Sirolimus: 20 mg/m2 every 2 weeks (28-day cycle) by IV.
  Modified FOLFOX6 regimen: oxaliplatin 85 mg/m2 IV with LV 400 mg/m2 IV over 2 hours plus FU 400 mg/m2 IV bolus and 2,400 mg/m2 continuous infusion over 46 hours every 2 weeks
  Bevacizumab: 5 mg/kg IV every 2 weeks
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Nab-Sirolimus 30 mg/m2 qw3/4 | Cohort 1: Nab-Sirolimus 20 mg/m2 qw3/4 | Cohort 2: Nab-Sirolimus 20 mg/m2 qw2/4 | Total
Number analyzed (Participants) | 6 | 10 | 44 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 9 | 34 | 47
  >=65 years | 2 | 1 | 10 | 13
Age, Continuous [Median (Full Range); unit: Years] | 61.5 [49 to 72] | 46.0 [34 to 71] | 51.0 [28 to 78] | 51.0 [28 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 17 | 23
  Male | 5 | 5 | 27 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 8 | 41 | 54
  Unknown or Not Reported | 1 | 2 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 0 | 1 | 3 | 4
  White | 6 | 7 | 36 | 49
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 6 | 10 | 44 | 60

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting-toxicities (DLTs) (Phase 1)
Description: Dose-limiting-toxicities within the first 2 cycles of treatment with nab-sirolimus at various doses and schedule in combination with mFOLFOX6 and bevacizumab
Time Frame: First 2 treatment cycles (2 months)
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Nab-Sirolimus 30 mg/m2 qw3/4: Dose / Schedule Cohort 1:
  nab-Sirolimus: 30 mg/m2 weekly on Days 1, 8, and 15 (28-day cycle) by IV
  Modified FOLFOX6 regimen: oxaliplatin 85 mg/m2 IV with LV 400 mg/m2 IV over 2 hours plus FU 400 mg/m2 IV bolus and 2,400 mg/m2 continuous infusion over 46 hours every 2 weeks
  Bevacizumab: 5 mg/kg IV every 2 weeks
- All Patients: The safety analysis set includes all treated patients
Arm/Group | Cohort 1: Nab-Sirolimus 30 mg/m2 qw3/4 | Cohort 2: Nab-Sirolimus 20 mg/m2 qw3/4 | Cohort 3: Nab-Sirolimus 20 mg/m2 qw2/4 | All Patients
Number analyzed (Participants) | 6 | 10 | 44 | 60
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Progression-free Survival at 6 Months (Phase 2) for All Patients, at the RP2D, as Well as Based on PTEN Status (Positive and Negative)
Description: The PFS rate at 6 months was estimated using the Kaplan-Meier method for a) all efficacy evaluable patients, b) patients receiving treatment at the RP2D, and c) based on PTEN status (positive or negative). Progression-free survival was defined as the time from the first day of study drug administration to disease progression or death due to any cause. Response evaluation was performed per RECIST v1.1, with the criteria for progression is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: 6 months
Population: The Efficacy Analysis Set includes all patients at baseline who received ≥2 doses of nab-sirolimus and had ≥1 scan. Based on the statistical design of this Phase 1/2 study, the efficacy endpoints are analyzed together for All Efficacy Evaluable patients (n=56) and at the RP2D (n=41). The data for all efficacy evaluable patients was also prospectively evaluated based on PTEN status for those with available IHC results (positive or negative, n=39 and n=12, respectively).
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- All Efficacy Evaluable Patients: The Efficacy Analysis Set includes all enrolled patients with measurable tumor per RECIST v1.1 at baseline who received at least 2 doses of ABI-009 and had a follow-up CT / PET (or MRI)
- RP2D (Cohort 3): Nab-Sirolimus 20 mg/m2 qw2/4: Dose / Schedule Cohort 3 (Recommended Phase 2 Dose, RP2D):
  nab-Sirolimus: 20 mg/m2 every 2 weeks (28-day cycle) by IV
  Modified FOLFOX6 regimen: oxaliplatin 85 mg/m2 IV with LV 400 mg/m2 IV over 2 hours plus FU 400 mg/m2 IV bolus and 2,400 mg/m2 continuous infusion over 46 hours every 2 weeks
  Bevacizumab: 5 mg/kg IV every 2 weeks
- PTEN Positive: PTEN positive patients in the Efficacy Analysis Set, regardless of dosing and schedule
- PTEN Negative: PTEN negative patients in the Efficacy Analysis Set, regardless of dosing and schedule
Arm/Group | All Efficacy Evaluable Patients | RP2D (Cohort 3): Nab-Sirolimus 20 mg/m2 qw2/4 | PTEN Positive | PTEN Negative
Number analyzed (Participants) | 56 | 41 | 39 | 12
percentage of patients | 77.3 [63.5 to 86.5] | 76.3 [59.2 to 86.9] | 78.2 [61.0 to 88.5] | 82.5 [46.1 to 95.3]

3. Secondary Outcome: Disease Control Rate (DCR) (Phase 2) for All Patients, at the RP2D, as Well as Based on PTEN Status (Positive and Negative)
Description: Disease control rate is defined as patients who achieved complete response, partial response, or stable disease and was summarized for a) all efficacy evaluable patients, b) patients receiving treatment at the RP2D, and c) based on PTEN status (positive or negative). Complete response and partial response required confirmation of response at the subsequent tumor assessment. Stable disease required a confirmatory assessment at a minimum interval of 8 weeks
Time Frame: Through study completion (up to 50 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of efficacy analysis patients
Groups:
- All Patients: The Efficacy Analysis Set includes all enrolled patients with measurable tumor per RECIST v1.1 at baseline who received at least 2 doses of ABI-009 and had a follow-up CT / PET (or MRI)
- RP2D (Cohort 3): Nab-Sirolimus 20 mg/m2 qw2/4: Dose / Schedule Cohort 3, (Recommended Phase 2 Dose, RP2D):
  nab-Sirolimus: 20 mg/m2 every 2 weeks (28-day cycle) by IV
  Modified FOLFOX6 regimen: oxaliplatin 85 mg/m2 IV with LV 400 mg/m2 IV over 2 hours plus FU 400 mg/m2 IV bolus and 2,400 mg/m2 continuous infusion over 46 hours every 2 weeks
  Bevacizumab: 5 mg/kg IV every 2 weeks
Arm/Group | All Patients | RP2D (Cohort 3): Nab-Sirolimus 20 mg/m2 qw2/4 | PTEN Positive | PTEN Negative
Number analyzed (Participants) | 56 | 41 | 39 | 12
percentage of efficacy analysis patients | 78.6 [65.6 to 88.4] | 75.6 [59.7 to 87.6] | 79.5 [63.5 to 90.7] | 83.3 [51.6 to 97.9]

4. Secondary Outcome: Median Progression-free Survival (Phase 2) for All Patients, at the RP2D, as Well as Based on PTEN Status (Positive and Negative)
Description: The median PFS was estimated using the Kaplan-Meier method for a) all efficacy evaluable patients, b) patients receiving treatment at the RP2D, and c) based on PTEN status (positive or negative). Progression-free survival was defined as the time from the first day of study drug administration to disease progression or death due to any cause. Response evaluation was performed per RECIST v1.1, with the criteria for progression is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: Through study completion (up to 50 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | All Patients | RP2D (Cohort 3): Nab-Sirolimus 20 mg/m2 qw2/4 | PTEN Positive | PTEN Negative
Number analyzed (Participants) | 56 | 41 | 39 | 12
Month | 10.9 [8.5 to 15.7] | 10.9 [7.3 to 14.5] | 13.1 [9.2 to 19.8] | 10.4 [5.5 to 22.4]

5. Secondary Outcome: Overall Response Rate (Phase 2) for All Patients, at the RP2D, as Well as Based on PTEN Status (Positive and Negative)
Description: The ORR was the proportion of patients who achieved a confirmed partial response or complete response per RECIST v1.1, and summarized for a) all efficacy evaluable patients, b) patients receiving treatment at the RP2D, and c) based on PTEN status (positive or negative). The ORR was reported along with exact 95% confidence intervals computed by the Clopper-Pearson method. Per RECIST v1.1, at each timepoint, objective tumor response for target lesions were assessed as such: Complete Response, disappearance of all target lesions, and pathological lymph nodes must have a reduction <10 mm; Partial Response, ≥30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Through study completion (up to 50 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of efficacy analysis patients
Arm/Group | All Patients | RP2D (Cohort 3): Nab-Sirolimus 20 mg/m2 qw2/4 | PTEN Positive | PTEN Negative
Number analyzed (Participants) | 56 | 41 | 39 | 12
percentage of efficacy analysis patients | 39.3 [26.5 to 53.2] | 36.6 [22.1 to 53.1] | 43.6 [27.8 to 60.4] | 41.7 [15.2 to 72.3]

ADVERSE EVENTS:
Time Frame: Safety and tolerability was monitored through continuous reporting of treatment-emergent and treatment-related AEs, Serious AEs, laboratory abnormalities, and incidence of patients experiencing dose modifications, dose delay/dose not given, and/or premature discontinuation of study drugs due to an AE. All AEs will be recorded by the investigator from the time the patient signs informed consent until 28 days after the last dose of study drugs (up to 50 months)
Groups:
- Cohort 2 Nab-Sirolimus 20 mg/m2 qw3/4: Dose / Schedule Cohort 2:
  nab-Sirolimus: 20 mg/m2 weekly on Days 1, 8, and 15 (28-day cycle) by IV
  Modified FOLFOX6 regimen: oxaliplatin 85 mg/m2 IV with LV 400 mg/m2 IV over 2 hours plus FU 400 mg/m2 IV bolus and 2,400 mg/m2 continuous infusion over 46 hours every 2 weeks
  Bevacizumab: 5 mg/kg IV every 2 weeks
- Total: The safety analysis set includes all treated patients
Arm/Group | Cohort 1: Nab-Sirolimus 30 mg/m2 qw3/4 | Cohort 2 Nab-Sirolimus 20 mg/m2 qw3/4 | Cohort 3: Nab-Sirolimus 20 mg/m2 qw2/4 | Total
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/10 | 3/44 | 4/60
Serious Adverse Events (participants affected / at risk) | 0/6 | 2/10 | 5/44 | 7/60
Other Adverse Events (participants affected / at risk) | 6/6 | 9/10 | 44/44 | 59/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Nab-Sirolimus 30 mg/m2 qw3/4 (N=6) | Cohort 2 Nab-Sirolimus 20 mg/m2 qw3/4 (N=10) | Cohort 3: Nab-Sirolimus 20 mg/m2 qw2/4 (N=44) | Total (N=60)
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Enterocolitis infectious (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Rectal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Nab-Sirolimus 30 mg/m2 qw3/4 (N=6) | Cohort 2 Nab-Sirolimus 20 mg/m2 qw3/4 (N=10) | Cohort 3: Nab-Sirolimus 20 mg/m2 qw2/4 (N=44) | Total (N=60)
Mucositis (Gastrointestinal disorders) | 4 | 5 | 31 | 40
Diarrhea (Gastrointestinal disorders) | 3 | 5 | 15 | 23
Nausea (Gastrointestinal disorders) | 1 | 5 | 15 | 21
Vomiting (Gastrointestinal disorders) | 1 | 2 | 8 | 11
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 3 | 7
Anal inflammation (Gastrointestinal disorders) | 0 | 0 | 5 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 4 | 5
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 4 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 2 | 3
Fatigue (General disorders) | 4 | 5 | 26 | 35
Mucosal inflammation (General disorders) | 1 | 3 | 9 | 13
Application site pain (General disorders) | 1 | 2 | 0 | 3
Oedema peripheral (General disorders) | 0 | 0 | 3 | 3
Myelossupression (Neutropenia) (Blood and lymphatic system disorders) | 4 | 5 | 9 | 18
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 3 | 14 | 17
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2 | 10 | 15
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 11 | 11
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2 | 5 | 9
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 | 1 | 6 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1 | 3 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 5 | 18 | 26
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1 | 8 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 3
Myelosuppression (Thrombocytopenia) (Blood and lymphatic system disorders) | 5 | 4 | 13 | 22
Myelosuppression (Anemia) (Blood and lymphatic system disorders) | 5 | 3 | 8 | 16
Weight decreased (Investigations) | 4 | 2 | 10 | 16
Lipase increased (Investigations) | 2 | 3 | 6 | 11
Amylase increased (Investigations) | 1 | 3 | 4 | 8
ALT (Investigations) | 0 | 0 | 5 | 5
AST (Investigations) | 0 | 0 | 5 | 5
Dysgeusia (Nervous system disorders) | 1 | 3 | 6 | 10
Headache (Nervous system disorders) | 0 | 2 | 4 | 6
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 3
Taste disorder (Nervous system disorders) | 1 | 1 | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 6 | 10
Infection (Infections and infestations) | 1 | 2 | 3 | 6
Candida infection (Infections and infestations) | 1 | 0 | 3 | 4
Hypoalbuminaemia (Hepatobiliary disorders) | 0 | 0 | 4 | 4
Proteinuria (Renal and urinary disorders) | 0 | 1 | 2 | 3
Dry eye (Eye disorders) | 0 | 0 | 3 | 3
Hypertension (Vascular disorders) | 0 | 1 | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 4 | 4
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT03439462/Prot_SAP_000.pdf